CLINICAL TRIAL: NCT04840329
Title: Endocation: A Randomized Cluster Controlled Trial of an Endometriosis Education Program for Middle and Secondary School Students
Brief Title: Endocation: Trial of an Endometriosis Education Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BC Women's Hospital & Health Centre (Other)
Collaborators: BC Support Unit (Other)
Responsible Party: Principal Investigator, Paul Yong, Associate Professor, BC Women's Hospital & Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: H19-00978
Record Dates: First submitted 2021-04-07; First posted 2021-04-12 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — Educational Status

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education Arm (Experimental)
  Interventions: Behavioral: Education
- Waitlist Control Arm (No Intervention)

INTERVENTIONS:
Behavioral: Education — One-time educational session about menstrual health and endometriosis
  Arms: Education Arm

SUMMARY:
Endometriosis is a common condition that affects 10% of females, causing chronic pain and other health concerns. Currently, it takes 8-12 years to be diagnosed with endometriosis, in part because there is low awareness of this condition. This research is designed to test whether providing endometriosis education in schools can help increase early awareness of the condition.

ELIGIBILITY:
Inclusion Criteria:

* 8-12 grade level class

Exclusion Criteria:

* Instruction offered in a language other than English

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2021-05-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline in menstrual health and endometriosis knowledge | Baseline and 4 weeks
  Assessed using a built for purpose questionnaire, possible scores range from 0 to 8

SECONDARY OUTCOMES:
Change from baseline in prioritization of menstrual health | Baseline and 4 weeks
  Assessed using a built for purpose item, possible scores range from 0 to 4
Change from baseline in confidence in endometriosis knowledge | Baseline and 4 weeks
  Assessed using a built for purpose item, possible scores range from 0 to 4
Change from baseline in comfort with menstrual health | Baseline and 4 weeks
  Assessed using a built for purpose item, possible scores range from 0 to 4
Acceptability of menstrual health and endometriosis education (quantitative) | Immediately following education in intervention and waitlist control group
  Assessed using a built for purpose questionnaire, possible scores range from 0 to 35
Acceptability of menstrual health and endometriosis education (qualitative) | Immediately following education in intervention and waitlist control group
  Assessed using open-ended responses a built for purpose questionnaire
Refusal of participants invited to participate | Baseline
  Number of participants who refuse to participate divided by the number of participants invited to participate
Retention of participants | 4 weeks
  Number of participants completing the study divided by the number of participants enrolled

CONTACTS AND LOCATIONS:
Overall Officials: Paul Yong, Principal Investigator — University of British Columbia
Locations (1):
- BC Women's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No